CLINICAL TRIAL: NCT04614480
Title: A Multicenter, Prospective, Multi-organ Study to Evaluate the Clinical Benefit of an Exome "Complex" Analysis Versus an Exome "Simple" Analysis to Help the Therapeutic Decision for the Precision Medicine
Brief Title: Exome Analysis (Complexe vs Simple) to Help the Therapeutic Decision for the Precision Medicine
Acronym: EXOMA2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A02135-52
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: genetic; exome
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Metastatic breast cancers (Other)
  Interventions: Genetic: Exome analysis
- Metastatic prostate cancers (Other)
  Interventions: Genetic: Exome analysis
- Metastatic lung cancers (Other)
  Interventions: Genetic: Exome analysis
- Metastatic colorectal cancers (Other)
  Interventions: Genetic: Exome analysis
- metastatic otorhinolaryngeal cancer (Other)
  Interventions: Genetic: Exome analysis
- metastatic ovarian cancer (Other)
  Interventions: Genetic: Exome analysis
- Pancreatic cancers (Other)
  Interventions: Genetic: Exome analysis
- Others metastatic cancers (Other)
  Interventions: Genetic: Exome analysis
- Metastatic sarcoma (Other)
  Interventions: Genetic: Exome analysis
- Metastatic gynecological cancer (Other)
  Interventions: Genetic: Exome analysis
- Metastatic renal cancer (Other)
  Interventions: Genetic: Exome analysis
- Metastatic cholangiocarcinoma metastatic (Other)
  Interventions: Genetic: Exome analysis
- Metastatic digestive cancer (other than stomach and colorectal) (Other)
  Interventions: Genetic: Exome analysis
- Metastatic stomach cancer (Other)
  Interventions: Genetic: Exome analysis

INTERVENTIONS:
Genetic: Exome analysis — Exome analysis of tumor DNA and constitutional DNA in patients included in 1st line treatment

SUMMARY:
The "simple" analysis of the exome can determine somatic and constitutional mutations. The major challenge lies in the translation of sequencing data into clinically relevant information allowing the clinician to guide his decision-making A "complex" analysis of the exome would provide access to structural DNA data, concerning mutational signatures, tumor mutational load, analysis of large deletions, loss of heterozygosity as well as amplification of certain genes which may have an impact on the management of patients.

No data available to date makes it possible to assess the clinical interest of the availability of its additional information resulting from a "complex" analysis compared to a "simple" analysis. The objective of the EXOMA2 study is to assess the proportion of patients for whom the proposed therapy is derived from its additional information (complex analysis) and would not have been possible with a classic exome analysis (simple analysis) .

We hereby formulate the hypothesis that a "complex" analysis on a population presenting a metastatic or locally advanced disease treated early (from the 1st line of treatment) will make it possible to determine therapeutic indications which could not be discovered with a "simple" analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Weight> 30 Kg
3. Histological or cytological evidence of the diagnosis of a metastatic or locally advanced solid tumor
4. Patient in 1st line of treatment for metastatic or locally advanced disease
5. Tumor material available in sufficient and usable quantity for the analyzes required by the study
6. Request for exome analysis to be carried out when initiating the 1st or 2nd line of treatment (line initiated at the time of inclusion)
7. Life expectancy estimated to be probably ≥ 6 months.
8. WHO ≤ 1
9. Patient capable and willing to follow all study procedures in accordance with the protocol
10. Patient having understood the purpose, risks and constraints of the study and having signed and dated the consent form
11. Patient affiliated to the social security scheme.

Exclusion Criteria:

1. Tumor material not available or biopsy not possible.
2. Inability to take a blood test.
3. Refusal of genetic analysis.
4. Patient likely to progress within 3 months of inclusion in the study.
5. History of HIV / HBV / HCV infection.
6. Patient already included in the EXOMA or EXOMA2 study.
7. Woman who is pregnant, may be, or is breastfeeding.
8. Persons deprived of their liberty or under guardianship (including curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7976 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2028-09-02 (Estimated); Study Completion 2032-09-02 (Estimated)

PRIMARY OUTCOMES:
proportion of patients for whom therapy was initiated from informations of the "complex" exome analysis | inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Charles Coutant, PU-PH, Study Director — Centre Georges François Leclerc
Locations (12):
- France (12):
  - CHU Amiens Picardie, Amiens
  - CHRU Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Henri Baclesse, Caen
  - CGFL, Dijon
  - CHU François Mitterrand, Dijon
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - CHU Nantes, Nantes
  - Chu Poitiers, Poitiers
  - Institut JeanGodinot, Reims
  - Centre Eugène Marquis, Rennes